CLINICAL TRIAL: NCT04526613
Title: A Cross-Sectional Study to Estimate the Influence of Malnutrition, Diabetes Mellitus and Helminth Infections on Biosignatures in Latent Tuberculosis in a South Indian Population
Brief Title: The Influence of Malnutrition, Diabetes Mellitus, and Helminth Infections on Biosignatures in Latent Tuberculosis in a South Indian Population
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920144; 20-I-N144
Record Dates: First submitted 2020-08-25; First posted 2020-08-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-03-27

CONDITIONS: Mycobacterium Tuberculosis; LTBI (Latent TB Infection); Malnutrition; Diabetes Mellitus; Helminth Infections
Keywords: MALNUTRITION; Diabetes Mellitus; Helminth Infections; Pathogenesis; Immunological Assays
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus; Trematode Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 'healthy' LTBI+ controls who are negative for all of the conditions: 'healthy' LTBI+ controls who are negative for all of the listed conditions
- healthy LTBI negative controls with none of the above conditio: healthy LTBI negative controls with none of the above conditions
- LTBI+ and helminth infection (positive stool qPCR and/or serol: LTBI+ and helminth infection (positive stool qPCR and/or serology)
- LTBI+ and severe to moderate malnutrition (BMI <17 kg/m2): LTBI+ and severe to moderate malnutrition (BMI <17 kg/m2)
- LTBI+ and uncontrolled DM (HbA1c >8%): LTBI+ and uncontrolled DM (HbA1c >8%)
- LTBI+ with more than one of the conditions defined in groups 1: LTBI+ with more than one of the conditions defined in groups 1-3

SUMMARY:
About 2 billion people worldwide are infected with tuberculosis (TB). Ninety percent of those people have latent TB infection (LTBI). Risk factors like malnutrition, diabetes mellitus (DM), and helminth infection can affect the development of active TB. Researchers want to study LTBI individuals with these issues to see how they may contribute to a person s higher risk for developing active TB. This study will take place in Chennai, India.

Objective:

To estimate the prevalence of malnutrition, DM, and helminth infections in people with LTBI.

Eligibility:

People age 14 65 with or without LTBI.

Design:

Participants will be screened with a medical history and physical exam focused on symptoms of active TB. Those who have TB symptoms will not take part in the study. Those who do not have TB symptoms will have a physical exam with vital signs, height, and weight. They will give blood and stool samples.

Participants will be assigned to 1 of 6 groups. They will repeat some of the screening tests. They will give urine samples. Some groups will have a chest X-ray. Some groups will have an ultrasound of the abdomen.

Participants will complete a survey about their history of smoking and drug and alcohol use.

Participants will have data collected about their nutritional status and body composition. Their skinfold thickness, ratio of waist/hip circumference, and grip strength will be measured.

Participants with DM, malnutrition, or helminth infection will be given standard of care or referred for follow-up treatment.

Participation will last up to 6 months.

...

DETAILED DESCRIPTION:
Approximately 2 billion people worldwide are infected with Mycobacterium tuberculosis (TB), with 90% of individuals having latent infection (LTBI). The control of TB requires clearly delineated helper T cell (Th) 1 responses and, to a lesser extent, Th17 responses, which both play important roles in the induction and maintenance of protective immune responses in mouse models of TB infection and in the prevention of active disease, as seen in LTBI. During latency, M. tuberculosis is contained in localized granulomas. Mycobacteria-specific T cells mediate delayed-type hypersensitivity reactions to purified protein derivative (PPD), and this reaction is generally considered to indicate an LTBI status in the absence of demonstrable active infection.

Among the various risk factors that are known to play a role in promoting active TB, HIV is the most well studied and described. However, in low-HIV-endemic countries like India, other risk factors might play a more prominent role in active TB pathogenesis. These include malnutrition, diabetes mellitus (DM), and helminth infections. LTBI individuals with these comorbidities or coinfections could be at a higher risk for developing active TB than their healthy LTBI counterparts without these comorbidities. Thus, it is imperative to study the pathogenesis of TB infection and disease in these at-risk populations.

In this study, we will estimate the prevalence of severe to moderate malnutrition, uncontrolled DM, and helminth infections in LTBI-positive individuals. We will collect samples from a cohort of individuals with LTBI, those with LTBI and coexistent malnutrition, DM, or helminth coinfection, and those without any of these conditions. Individual participation may last up to 6 months. The main objective of the study is to estimate the prevalence of malnutrition, DM, and helminth infections in LTBI individuals.

Simultaneously, we will perform transcriptomic, proteomic, and metabolomic assays, including profiles in serum and urine, to determine the biosignature portfolio of these individuals. In addition, immunological assays examining cytokine/chemokine signatures as well as other immune parameters related to innate and adaptive responses will be performed to enhance the understanding of the immunological cross-talk between LTBI and malnutrition, DM, and helminth infections.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA (Screening Phase)

Individuals who meet the following criteria are eligible to participate in the screening phase:

* Aged 14 to 65 years.
* Willingness to provide blood, urine, and stool samples for examination.
* Willingness to have samples and data stored.
* Able to provide informed consent.

PARTICIPANT EXCLUSION CRITERIA (Screening Phase)

* Pulmonary symptoms suggestive of TB (cough >2 weeks in duration and/or intermittent fever >1 week in duration and/or hemoptysis).
* Two IGRA tests with indeterminate results (mitogen values <10 IU).

PARTICIPANT INCLUSION CRITERIA (Study Phase)

Individuals are eligible for the study phase if they meet the requirements for one of the study groups, as follows:

1. LTBI+ and severe to moderate malnutrition (BMI <17 kg/m2);
2. LTBI+ and uncontrolled DM (HbA1c >8%);
3. LTBI+ and helminth infection (positive stool qPCR and/or serology);
4. LTBI+ with more than one of the conditions defined in groups 1 3;
5. healthy LTBI+ controls who are negative for all of the above conditions; and
6. healthy LTBI-negative controls with none of the above conditions.

PARTICIPANT EXCLUSION CRITERIA (Study Phase)

* Pulmonary symptoms suggestive of TB (cough >2 weeks in duration and/or intermittent fever >1 week in duration and/or hemoptysis).
* Pregnant or lactating women.
* Previous treatment for LTBI.
* Anemia with hemoglobin <8 g/dl (evaluated at the screening phase visit).
* For LTBI+ participants, clinically indicated chest X-ray positive for pulmonary TB.
* For malnourished participants, clinically indicated abdominal ultrasound positive for abdominal TB.
* Known documented cases of cancer, acquired immune deficiency syndrome, or other immunosuppressive illness.
* History of any other illness or condition which, in the investigator s judgment, may substantially increase the risk associated with the participant s participation in the protocol, or compromise the scientific objectives.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from villages in the Kancheepuram District in south India. The census in villages in the Kancheepuram District is updated annually by local health workers employed by the Department of Public Health and the field teams of the NIRT in Chennai, India. The villages will be chosen in consultation with the Department of Public Health in Tamil Nadu.
Sampling Method: Non-Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malnutrition, DM and helminth infections in LTBI individuals and their effects on biosignatures | Study Phase visit
  Prevalence of malnutrition, DM and helminth infections in LTBI individuals and their effects on biosignatures

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute for Research In Tuberculosis, International Centers for Exel, Chennai, India

IPD SHARING:
Plan to Share IPD: No
This is a sample/data collection study to estimate the prevalence of malnutrition. DM and helminth infections in LBTI subjects. There is no plan to share individual participant data

REFERENCES:
- [Background] Barry CE 3rd, Boshoff HI, Dartois V, Dick T, Ehrt S, Flynn J, Schnappinger D, Wilkinson RJ, Young D. The spectrum of latent tuberculosis: rethinking the biology and intervention strategies. Nat Rev Microbiol. 2009 Dec;7(12):845-55. doi: 10.1038/nrmicro2236. Epub 2009 Oct 26. PMID 19855401
- [Background] Lin PL, Flynn JL. Understanding latent tuberculosis: a moving target. J Immunol. 2010 Jul 1;185(1):15-22. doi: 10.4049/jimmunol.0903856. PMID 20562268